CLINICAL TRIAL: NCT03079466
Title: Effect of CPAP Treatment on the Elderly With Mild to Moderate Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitario Doctor Peset (Other)
Responsible Party: Principal Investigator, Silvia Ponce Perez, Doctor, Hospital Universitario Doctor Peset
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sleep workgroup
Record Dates: First submitted 2017-03-09; First posted 2017-03-14 (Actual); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Unrecognized Condition
Keywords: Sleep apnea; Elderly; CPAP
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment CPAP (Active Comparator): A group treated with CPAP
  Interventions: Other: CPAP
- group without treatment (Sham Comparator)
  Interventions: Other: CPAP

INTERVENTIONS:
Other: CPAP — This is a randomized study where patients are included consecutively under a randomization order that will be given to the investigators. Patients will continue to be treated with CPAP and other treatment with no CPAP for a duration of 3 months and with intention-to-treat analysis And by protocol.

SUMMARY:
Objective: To analyze the impact of CPAP treatment on cognitive, clinical and quality of life domains in patients over 70 years of age with mild-to-moderate OSA

Primary Outcome: Epworth scale and QSQ domains

Secondary Outcomes: Neurocognitive variables and CPAP adherence

ELIGIBILITY:
Inclusion Criteria:

* Age equal or greater than 70 years of both sexes
* Patients with sleep study results with AHI ≥ 15 and < 30

Exclusion Criteria:

* Alternative diagnoses of other non-respiratory sleep disorders that are also cause of pathological somnolence (eg, sdr restless legs, narcolepsy, etc.)
* Don't sign informed consent
* Acute or chronic respiratory insufficiency requiring home oxygen therapy
* Patients with Obesity Hypoventilation Syndrome
* Diagnosis of neuro-psychiatric diseases with the exception of anxiety - depression or diagnosis of dementia.
* Diseases of any origin in the acute phase
* Heart failure or recent stroke (less than 3 months).
* Central SAHS (more than 50% of the registry with central apneas or Cheyne-Stokes breathing)
* Pre-treatment with CPAP
* Inability to perform the diagnostic study of sleep due to the patient's condition
* Hipersomniaincapacitante (Epworth≥18) with no known or most likely cause related to SAHS

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2017-06-10 (Estimated); Study Completion 2017-07-15 (Estimated)

PRIMARY OUTCOMES:
Epworth Sleepiness Scale | 3 months
  Measure of diurnal sleepiness
Quebec Sleep Questionnaire domains | 3 months
  Quality of Life measured in sleep apnea patients

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Martinez-Garcia MA, Oscullo G, Ponce S, Pastor E, Orosa B, Catalan P, Martinez A, Hernandez L, Muriel A, Chiner E, Vigil L, Carmona C, Mayos M, Garcia-Ortega A, Gomez-Olivas JD, Beauperthuy T, Bekki A, Gozal D. Effect of continuous positive airway pressure in very elderly with moderate-to-severe obstructive sleep apnea pooled results from two multicenter randomized controlled trials. Sleep Med. 2022 Jan;89:71-77. doi: 10.1016/j.sleep.2021.11.009. Epub 2021 Nov 24. PMID 34915264